CLINICAL TRIAL: NCT00517309
Title: Immunogenicity and Safety of Quadrivalent HPV L1 Virus-Like Particle (VLP) Vaccine in 16- to 23-Year-Old Women When Administered Alone or Concomitantly With Hepatitis B Vaccine (Recombinant)--the F.U.T.U.R.E. Study (Females United to Unilaterally Reduce Endo/Ectocervical Disease
Brief Title: Study to Test the Safety of HPV Vaccine in Women (V501-011)(COMPLETED)
Acronym: FUTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-011; 2007_576
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Cervical Cancer; Genital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Vaccines, Synthetic; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Biological: V501, Gardasil, Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine / Duration of Treatment : 4 Years
Biological: Comparator: placebo (concomitant-vaccine matched) / Duration of Treatment : 4 Years

SUMMARY:
The primary purpose of the study is to test the safety of HPV Vaccine in Women

ELIGIBILITY:
Inclusion Criteria:

* Females age 16 to 23 years old
* Must agree to refrain from sexual activity (vaginal or anal) for 48 hours prior to any scheduled visit

Exclusion Criteria:

* History of vaccination with an HPV vaccine
* History of hepatitis B infection
* History of vaccination with hepatitis B vaccine
* History of genital warts or treatment for genital warts

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1877 (Actual)
Dates: Start 2001-12-28 (Actual); Primary Completion 2004-06-08 (Actual); Study Completion 2004-06-11 (Actual)

PRIMARY OUTCOMES:
Quadrivalent HPV vaccine is generally well tolerated when administered alone or concomitantly with hepatitis B vaccine.

SECONDARY OUTCOMES:
HPV vaccine is well tolerated in 16-23 year old females.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Wheeler CM, Bautista OM, Tomassini JE, Nelson M, Sattler CA, Barr E; Protocol 11 study Investigators. Safety and immunogenicity of co-administered quadrivalent human papillomavirus (HPV)-6/11/16/18 L1 virus-like particle (VLP) and hepatitis B (HBV) vaccines. Vaccine. 2008 Jan 30;26(5):686-96. doi: 10.1016/j.vaccine.2007.11.043. Epub 2007 Dec 5. PMID 18164106
- [Background] Giuliano AR, Lazcano-Ponce E, Villa L, Nolan T, Marchant C, Radley D, Golm G, McCarroll K, Yu J, Esser MT, Vuocolo SC, Barr E. Impact of baseline covariates on the immunogenicity of a quadrivalent (types 6, 11, 16, and 18) human papillomavirus virus-like-particle vaccine. J Infect Dis. 2007 Oct 15;196(8):1153-62. doi: 10.1086/521679. Epub 2007 Sep 17. PMID 17955433
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html